CLINICAL TRIAL: NCT06744192
Title: A Prospective Case-control Clinical Study of the Ultrasound Imaging Reporting and Data System for Diagnosis of Anterosuperior Acetabular Labral Tears
Status: Completed | Type: Observational
Sponsor: Yi Mao (Other)
Responsible Party: Sponsor-Investigator, Yi Mao, Postgraduate Student, and Research Assistant in Ultrasound Department, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: ChinaPLAGH202412
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Acetabular Labrum Tear; Ultrasound Exams; Diagnostic Imaging; Models

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — This study was a non-invasive imaging examination and did not involve sample acquisition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- tear: Patients diagnosed hip labrum tear by a hip arthroscopy or by a comprehensive clinical diagnosis through an orthopaedic surgeon with 15 years of experience
- non-tear: Patients no diagnosed hip labrum tear by a hip arthroscopy or by a comprehensive clinical diagnosis through an orthopaedic surgeon with 15 years of experience

SUMMARY:
The goal of this clinical trial is to develop an ultrasonic imaging reporting and data system for diagnosis of anterosuperior acetabular labral tears (ALT). Participants will receive a comprehensive clinical diagnosis or a hip arthroscopy to determine whether there is a torn labrum of the hip. Comparing the ultrasonographic characteristics of hip labrum in tear group and non-tear group, establishing diagnostic model is conducive to early diagnosis and differential diagnosis of this disease.

ELIGIBILITY:
Inclusion criteria: a)18 years of age and above; b) Combined with clinical symptoms, signs, and MRI, a senior orthopaedic surgeon or a final arthroscopy will determine whether the labrum of the hip is torn.

Exclusion criteria: a) other diseases affecting the hip joint (tumors, infections and fractures); b) A history of hip surgery; c)BMI≥30 kg/m²; d) Pregnant patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the First Medical Center and the Fourth Medical Center of the PLA General Hospital included patients with orthopedic hip discomfort and patients admitted to the ultrasound department without hip injury.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
labral echo homogeneity | After the completion of data collection and a week of data collation, two ultrasound physicians who had undergone one month of specialized reading training spent two weeks interpreting the hip labrum ultrasound images of all participants.
  Labral echo homogeneity is divided into homogeneous and heterogeneous.
labral shape | After the completion of data collection and a week of data collation, two ultrasound physicians who had undergone one month of specialized reading training spent two weeks interpreting the hip labrum ultrasound images of all participants.
  Labral shape was divided into regular and irregular (there are potholes at the lip edge of the labrum or labrum are too full and swollen).
labral hypoechoic cleft | After the completion of data collection and a week of data collation, two ultrasound physicians who had undergone one month of specialized reading training spent two weeks interpreting the hip labrum ultrasound images of all participants.
  Whether to tear was divided into yes and no.
labral focal hyperechoic area | After the completion of data collection and a week of data collation, two ultrasound physicians who had undergone one month of specialized reading training spent two weeks interpreting the hip labrum ultrasound images of all participants.
  According to whether there is a focal hyperechoic area in the acetabular labrum, it is divided into yes and no.
labral echogenicity | After the completion of data collection and a week of data collation, two ultrasound physicians who had undergone one month of specialized reading training spent two weeks interpreting the hip labrum ultrasound images of all participants.
  Echo intensity can be divided into Hypoecho, Isoecho and hyperecho.
Paralabral cysts | After the completion of data collection and a week of data collation, two ultrasound physicians who had undergone one month of specialized reading training spent two weeks interpreting the hip labrum ultrasound images of all participants.
  Absent or Present
Cortical Bone of Ilium | After the completion of data collection and a week of data collation, two ultrasound physicians who had undergone one month of specialized reading training spent two weeks interpreting the hip labrum ultrasound images of all participants.
  According to the continuity of the cortical bone of the ilium, it can be divided into continuous and interrupted.
Max cross-section area of labrum | After the data collection and a week of data collation, two ultrasound physicians undergone one month of specialized reading training spent two weeks interpreting the hip labrum ultrasound of all participants. Take the average value of three times.
  The largest area of the anterior superior labrum of the hip.
Hip Capsule Thickness | After the data collection and a week of data collation, two ultrasound physicians undergone one month of specialized reading training spent two weeks interpreting the hip labrum ultrasound of all participants. Take the average value of three times.
  The anterior superior articular capsule of the hip was ultrasonically measured in the thickest area.
Thickness of Articular Cavity | n and a week of data collation, two ultrasound physicians undergone one month of specialized reading training spent two weeks interpreting the hip labrum ultrasound of all participants. Take the average value of three times.
  The ultrasound was located at the longitudinal section of the femoral neck and measured the maximum thickness of the joint cavity of the femoral neck recess.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Medical Center of the PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No